CLINICAL TRIAL: NCT05446974
Title: Development of Training Programs for Nursing Competency Reinforcement to Spread Trauma Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4-2021-0324
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Nurses Who Work at the Community Mental Health Welfare Center

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing intervention (Experimental): Nurses randomly assigned by applying a random selection method
  Interventions: Other: Nursing Competency Enhancement Training Program in PTSD Intervention
- Non-intervention (No Intervention): Nurses randomly assigned by applying a random selection method

INTERVENTIONS:
Other: Nursing Competency Enhancement Training Program in PTSD Intervention — This program was for nurses who work at the Mental Health Welfare Center and consisted of a workbook, self-learning online education, and workshop. It included a spoken audio track that was accompanied by visual prompts to provide knowledge on traumatic stress and introduce trauma recovery methods. Its online format made it convenient and widely accessible, and allowed for a low-intensity, cost-effective educational program. The program focused on providing self-learning guidelines for nurses to develop their capacity for PTSD intervention.
  Arms: Nursing intervention

SUMMARY:
This study aims to improve the trauma intervention competency of nurses through online-based training of the nursing intervention program for trauma-experienced subjects. The specific goals are as follows.

1. Based on Swanson's Caring Theory, develop an online training program for nurses to spread trauma nursing intervention and improve competency.
2. Evaluate the effects of the developed program's workbook and online training on nurses' trauma-related knowledge and attitude, self-efficacy, and professional quality of life.

Of the 42 subjects who enrolled in the study, 1 dropped out before intervention, resulting in 41 participants who completed all interventions and surveys.

ELIGIBILITY:
Inclusion Criteria:

* Those who have a nurse's license
* Those who work at the Mental Health Welfare Center
* Those who can access the program through a computer or mobile
* Those who understand the purpose of the research and voluntarily agree to participate in the research

Exclusion Criteria:

- Those who do not agree to participate in the study

Ages: 23 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Attitudes and knowledge about PTSD | one month after the intervention
  Attitudes and knowledge about PTSD; K-PTSD was used for attitudes and knowledge about PTSD.
  The attitude towards PTSD consists of 8 items, 5 items on attitude toward government policy and 3 items on attitude towards PTSD patients, and is evaluated on a 4-point scale.
  The general knowledge about PTSD consists of 8 questions, and the answer is very much (1 point), somewhat like it (2 points), not at all (3 points), and not at all (4 points). The range is 0 to 8 points. The knowledge about treatment consists of three questions, and it is a multiple choice type, and only one answer is correct, so the percentage of correct answers can be obtained.
Pro QOL | one month after the intervention
  Pro QOL: To measure the quality of life of experts, the Korean version of the Quality of Life Scale (K-ProQOL 5), which was validated by mental health experts, was used. It consists of a total of 30 questions and is evaluated on a 5-point scale. Sub-domains are divided into empathic satisfaction, exhaustion, and indirect trauma stress. A higher score means a higher level of each domain. Classification according to the cut-off point is divided into high, average, and low, and in the case of empathy satisfaction, 30 points or less means low, 31-37 points mean average, and 38 points or more means high. In the case of burnout, 20 points or less means low, 21-27 points mean average, and 28 points or more means good. Indirect trauma stress 18 or less, 19-25 points average, 26 or more means good .
Self efficacy | one month after the intervention
  Self efficacy: In order to measure the self-efficacy related to trauma intervention, the items developed for measuring confidence and perception related to trauma work were translated into Korean. It consists of a total of 12 items, and the perception of trauma-related task performance, work confidence, knowledge and skills is divided into five items on a 10-point scale (0: not at all, 10: very high). was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim S, Kim GU, Park J. Evaluation of Internet-Based Training in Trauma Care for Nurses in Mental Health Welfare Centers: A Cluster Randomized Controlled Trial. J Prim Care Community Health. 2023 Jan-Dec;14:21501319231181982. doi: 10.1177/21501319231181982. PMID 37335037